CLINICAL TRIAL: NCT01712230
Title: Bioenergetic and Metabolic Consequences of the Loss of Ovarian Function in Women
Brief Title: Females, Aging, Metabolism, and Exercise
Acronym: FAME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 12-1157; P50HD073063 (NIH)
Record Dates: First submitted 2012-10-19; First posted 2012-10-23 (Estimated); Results first posted 2019-11-22 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Obesity
Keywords: hormone therapy; obesity; menopause; disease /disorder proneness /risk; insulin sensitivity /resistance; metabolic syndrome; women's health
MeSH Terms: conditions — Obesity; Disease Susceptibility; Metabolic Syndrome | interventions — Gonadotropin-Releasing Hormone; Leuprolide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Monthly placebo injections for 6 months
  Interventions: Drug: Placebo
- GnRH agonist (Active Comparator): Monthly GnRH agonist injections for 6 months
  Interventions: Drug: GnRH agonist
- GnRH agonist + exercise (Active Comparator): Monthly GnRH agonist injections for 6 months plus supervised cardiovascular exercise intervention
  Interventions: Drug: GnRH agonist; Behavioral: Supervised cardiovascular exercise

INTERVENTIONS:
Drug: GnRH agonist — Drug: leuprolide acetate
  Other Names:
  Lupron 3.75 mg for depot suspension delivered by monthly intramuscular injection for 6 months
  Other Names: Leuprolide Acetate 3.75mg
  Arms: GnRH agonist; GnRH agonist + exercise
Behavioral: Supervised cardiovascular exercise — Supervised exercise, 4 days per week for 45 to 60 minutes per session for 6 months
  Arms: GnRH agonist + exercise
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study is designed to determine whether a reduction in hormones (such as occurs during menopause) causes a decrease in calories burned during physical activity. This study will also determine whether a reduction in hormones decreases calories burned while sleeping, resting, and eating and whether an exercise intervention can prevent this.

DETAILED DESCRIPTION:
Participants will be women who are nearing menopause based on age (42-52 y) but have normal menstrual cycles. Participants will be randomized to receive monthly injections of placebo or a study drug that reduces sex hormones (GnRH agonist) for 24 weeks. Women who receive GnRH agonist will be further randomized to no exercise or a supervised exercise program. Thus, the 3 treatment groups are: placebo, GnRH agonist, GnRH agonist+exercise. The investigators will measure changes in calories burned during physical activity, sleep, rest, and after a meal after 3 and 6 months of hormone suppression using doubly-labeled water and room calorimetry. Other measures include food intake estimated from food records; body composition measured by dual-energy x-ray absorptiometry (DXA); glucose and insulin responses to an oral glucose tolerance test; and markers of inflammation in the blood.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy women aged 40 to 60 years
2. Are still experiencing regular menstrual cycles.
3. They must be willing to be randomized to placebo or GnRHAG therapy for 24 weeks
4. Be physically able to be randomized to participate in a programmed exercise training program.

The investigators will consent up to 132 subjects with the aim of enrolling 22 in each of the 3 groups (placebo, GnRHAG, or GnRHAG+Exercise).

Exclusion Criteria:

* irregular menstrual cycles defined as 2 or more missed cycles in the previous year
* serum FSH >25 mIU/mL measured during the first 5 days of the menstrual cycle
* on hormonal contraceptive or menopausal therapy
* positive pregnancy test
* intention to become pregnant or start hormonal contraceptive therapy during the period of study
* lactation
* known hypersensitivity to GnRH or leuprolide acetate
* score >16 on the CESD((Center for Epidemiologic Studies Depression Scale )
* severe osteopenia or osteoporosis (i.e., proximal femur or lumbar spine t scores < -2.0)
* abnormal vaginal bleeding
* thyroid dysfunction, defined as an ultrasensitive TSH <0.5 or >5.0 mU/L; volunteers with abnormal TSH values will be re-considered for participation in the study after follow-up evaluation by the PCP with initiation or adjustment of thyroid hormone replacement
* uncontrolled hypertension defined as resting systolic BP >150 mmHg or diastolic BP>90 mmHg; participants who do not meet these criteria at first screening will be re-evaluated, including after follow-up evaluation by the PCP with initiation or adjustment of anti-hypertensive medications
* cardiovascular disease; subjective or objective indicators of ischemic heart disease (e.g., angina, ST segment depression) or serious arrhythmias at rest or during the graded exercise test (GXT) without follow-up evaluation; follow-up evaluation must include diagnostic testing (e.g., thallium stress test) with interpretation by a cardiologist
* orthopedic or other problems that would interfere with participation in the exercise program
* exercising at least 30 minutes per day at a moderate to vigorous intensity most days of the week (defined as >4 d/wk) over the past 6 months
* BMI <40 kg/m2

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2012-10; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Kohrt, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado - Anschutz Medical Campus, Aurora, Colorado, United States

REFERENCES:
- [Derived] Gavin KM, Melanson EL, Hildreth KL, Gibbons E, Bessesen DH, Kohrt WM. A Randomized Controlled Trial of Ovarian Suppression in Premenopausal Women: No Change in Free-Living Energy Expenditure. Obesity (Silver Spring). 2020 Nov;28(11):2125-2133. doi: 10.1002/oby.22978. PMID 33150745

RESULTS

PARTICIPANT FLOW:
Groups:
- GnRH Agonist: Monthly GnRH agonist injections for 6 months
  GnRH agonist: Drug: leuprolide acetate
  Other Names:
  Lupron 3.75 mg for depot suspension delivered by monthly intramuscular injection for 6 months
- GnRH Agonist + Exercise: Monthly GnRH agonist injections for 6 months plus supervised cardiovascular exercise intervention
  GnRH agonist: Drug: leuprolide acetate
  Other Names:
  Lupron 3.75 mg for depot suspension delivered by monthly intramuscular injection for 6 months
  Supervised cardiovascular exercise: Supervised exercise, 4 days per week for 45 to 60 minutes per session for 6 months
Period: Overall Study
Arm/Group | Placebo | GnRH Agonist | GnRH Agonist + Exercise
Started | 11 | 18 | 18
Completed | 9 | 14 | 11
Not Completed | 2 | 4 | 7

BASELINE CHARACTERISTICS:
Population: 47 women were enrolled in to the study, but only 42 completed the intervention. Baseline characteristics are reported for these 42 women. Primary and secondary outcome analyses were completed on 34 women who met the definition of compliance to the intervention (defined as completing >70% of prescribed exercise sessions).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | GnRH Agonist | GnRH Agonist + Exercise | Total
Number analyzed (Participants) | 10 | 14 | 18 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (1.7) | 47.1 (3.7) | 45.7 (3.0) | 46.3 (3.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 14 | 18 | 42
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 3 | 8
  Not Hispanic or Latino | 7 | 11 | 15 | 33
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 1 | 6
  White | 5 | 11 | 16 | 32
  More than one race | 2 | 1 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0
Physical Activity Energy Expenditure (PAEE) [Mean (Standard Deviation); unit: kcal/day] — PAEE is calculated as: TEE - REE - TEF, where TEE is total energy expenditure (measured by doubly-labeled water), REE is resting energy expenditure (measured by indirect calorimetry), and TEF is the thermic effect of feeding (estimated using a constant).
  kcal/day | 610 (315) | 630 (217) | 737 (295) | 671 (276)

OUTCOME MEASURES:

1. Primary Outcome: Change in Physical Activity Energy Expenditure (PAEE)
Description: PAEE will be calculated as: TEE - REE - TEF, where TEE is total energy expenditure (measured by doubly-labeled water), REE is resting energy expenditure (measured by indirect calorimetry), and TEF is the thermic effect of feeding (estimated using a constant).
Time Frame: Change from baseline to 6 months
Population: Placebo: One participant dropped because they got a new job. GnRH agonist+exercise: One participant dropped because of a health problem unrelated to the study. Results from five participants were not included in the analysis because they did not meet the exercise compliance threshold (completed <70% of exercise sessions).
Measure: Mean (Standard Error); unit: kcal/day
Arm/Group | Placebo | GnRH Agonist | GnRH Agonist + Exercise
Number analyzed (Participants) | 9 | 14 | 11
kcal/day | 74.5 (77.9) | -10.2 (63.6) | 61.0 (66.4)

2. Secondary Outcome: Total Fat Mass
Description: Total Fat mass as measured by DXA
Time Frame: Change over 6 months
Measure: Mean (Standard Error); unit: kg
Arm/Group | Placebo | GnRH Agonist | GnRH Agonist + Exercise
Number analyzed (Participants) | 9 | 14 | 11
kg | 0.73 (0.68) | 1.66 (0.41) | 0.89 (0.60)

3. Secondary Outcome: Total Fat Free Mass
Description: Total Fat Free Mass as measured by DXA
Time Frame: Change over 6 months
Measure: Mean (Standard Error); unit: kg
Arm/Group | Placebo | GnRH Agonist | GnRH Agonist + Exercise
Number analyzed (Participants) | 9 | 14 | 11
kg | 0.1 (0.34) | -0.69 (0.34) | -0.66 (0.59)

ADVERSE EVENTS:
Time Frame: 6 Months
Arm/Group | Placebo | GnRH Agonist | GnRH Agonist + Exercise
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/14 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/14 | 0/18
Other Adverse Events (participants affected / at risk) | 3/10 | 4/14 | 4/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | GnRH Agonist (N=14) | GnRH Agonist + Exercise (N=18)
Nausea/vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness/Hot Flash (Endocrine disorders) | 1 (1) | 0 (0) | 2 (2)
Bruising/tenderness from study procedure (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Mental state change (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) — Anxiety and decrease in perceived metal sharpness
Migraine (General disorders) | 1 (1) | 2 (2) | 0 (0)
Hamstring cramping (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vaginal bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Itching/blistering (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Itching/blistering of skin after tegaderm use

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-15): https://cdn.clinicaltrials.gov/large-docs/30/NCT01712230/Prot_SAP_000.pdf